CLINICAL TRIAL: NCT04661579
Title: A Phase 2b Randomized, Open-label, Controlled, Single Center Study in Plasmodium Falciparum-infected and Uninfected Adults Age 18-55 Years Old in Kenya to Evaluate the Efficacy of the Delayed, Fractional Dose RTS,S/AS01E Malaria Vaccine in Subjects Treated With Artemisinin Combination Therapy Plus Primaquine
Brief Title: Study of Malaria Vaccine RTS,S/AS01E in Plasmodium Falciparum-infected and Uninfected Adults Pre-treated With Anti-malarial Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry); Kenya Medical Research Institute (Other); FHI Clinical SA Proprietary Limited (Industry); DF/Net (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CVIA 078; PACTR202006896481432 (Registry Identifier: Pan African Clinical Trial Registry)
Record Dates: First submitted 2020-10-26; First posted 2020-12-10 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-01

CONDITIONS: Plasmodium Falciparum
Keywords: RTS,S/AS01E; hypo-immuno-responsiveness; open-label randomized study; Phase 2b; Kenyan adults; anti-malarials; fractional dose RTS,S/AS01E
MeSH Terms: conditions — Malaria, Falciparum | interventions — RTS malaria vaccine; Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Intervention Model Description: Three groups (Groups 1, 2, and 3) will be administered RTS,S/AS01E on a 0, 1, 7 month schedule with Dose 3 delivered as a 1/5th fractional dose. Two groups (Groups 4 and 5) will be administered a comparator vaccine on a 0, 1, 7 month schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Positive Parasitemia; Anti-malarial treatment + RTS,S/AS01E Vaccine (Experimental): Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with dihydroartemisinin-piperaquine (DHA/Pip) plus low dose primaquine (LD PQ) 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a course of artemether/lumefantrine (A/L) plus LD PQ was administered.
  Participants received 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
  Interventions: Biological: Malaria Vaccine RTS,S/AS01E; Drug: Dihydroartemisinin-piperaquine (DHA/Pip); Drug: Artemether / Lumefantrine; Drug: Primaquine
- Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine (Experimental): Participants with no detectable P. falciparum parasitemia at baseline received anti-malarial prophylaxis with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and a 2nd course of DHA/Pip plus LD PQ 2 weeks before the second vaccination. One week before the third vaccination, a course of A/L plus LD PQ was administered.
  Participants received 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
  Interventions: Biological: Malaria Vaccine RTS,S/AS01E; Drug: Dihydroartemisinin-piperaquine (DHA/Pip); Drug: Artemether / Lumefantrine; Drug: Primaquine
- Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine (Experimental): Participants with detectable P. falciparum parasitemia at baseline did not receive any anti-malarial medications to clear parasites.
  Participants received 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
  This group is included only for immunological assessment and not for vaccine efficacy.
  Interventions: Biological: Malaria Vaccine RTS,S/AS01E
- Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine (Placebo Comparator): Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with dihydroartemisinin-piperaquine (DHA/Pip) plus low dose primaquine (LD PQ) 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a three-day course of artemether/lumefantrine (A/L) plus LD PQ was administered.
  Participants received 3 vaccinations of Abhayrab rabies vaccine on a 0, 1, 7 month schedule.
  Interventions: Biological: Abhayrab rabies vaccine; Drug: Dihydroartemisinin-piperaquine (DHA/Pip); Drug: Artemether / Lumefantrine; Drug: Primaquine
- Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine (Placebo Comparator): Participants with no detectable P. falciparum parasitemia at baseline received anti-malarial prophylaxis with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and a 2nd course of DHA/Pip plus LD PQ 2 weeks before the second vaccination. One week before the third vaccination, a course of A/L plus LD PQ was administered.
  Participants received 3 vaccinations of Abhayrab rabies vaccine on a 0, 1, 7 month schedule.
  Interventions: Biological: Abhayrab rabies vaccine; Drug: Dihydroartemisinin-piperaquine (DHA/Pip); Drug: Artemether / Lumefantrine; Drug: Primaquine

INTERVENTIONS:
Biological: Malaria Vaccine RTS,S/AS01E — RTS,S/AS01E vaccine 0.5 mL, containing 25 μg protein comprising circumsporozoite protein (CS) and hepatitis B surface antigen (RTS,S), 25 μg monophosphoryl lipid (AMPL), 25 μg Quillaja saponaria 21 (QS21) in a liposomal formulation) for the first two immunizations. One-fifth dose RTS,S/AS01E vaccine was used for the third immunization.
  Arms: Group 1: Positive Parasitemia; Anti-malarial treatment + RTS,S/AS01E Vaccine; Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine; Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine
Biological: Abhayrab rabies vaccine — Abhayrab rabies vaccine, 0.5 mL, contains 2.5 IU rabies antigen.
  Arms: Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine; Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Drug: Dihydroartemisinin-piperaquine (DHA/Pip) — Dihydroartemisinin (120 mg or 160 mg based on weight) and piperaquine tetraphosphate (960 mg or 1280 mg based on weight) mg) administered once a day for 3 days.
  DHA/Pip is a long acting anti-malarial used to clear asexual stage and young gametocyte parasites.
  Arms: Group 1: Positive Parasitemia; Anti-malarial treatment + RTS,S/AS01E Vaccine; Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine; Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine; Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Drug: Artemether / Lumefantrine — Artemether (80 mg) and lumefantrine (480 mg) administered twice a day for 3 days.
  Coartem is a short-acting artemisinin combination therapy used to provide clearance of blood stage parasites in order to establish a clean baseline for determination of vaccine efficacy.
  Other Names: Coartem®
  Arms: Group 1: Positive Parasitemia; Anti-malarial treatment + RTS,S/AS01E Vaccine; Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine; Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine; Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Drug: Primaquine — One dose of 15 mg primaquine. Low dose primaquine (LD PQ) is used to clear mature gametocytes of P. falciparum.
  Arms: Group 1: Positive Parasitemia; Anti-malarial treatment + RTS,S/AS01E Vaccine; Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine; Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine; Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine

SUMMARY:
The main goal of this study is to assess the efficacy of RTS,S/AS01E, a candidate vaccine against malaria caused by Plasmodium falciparum (P. falciparum), in adults positive for P. falciparum at the start of the study, but treated with anti-malarial medications to clear the parasite before receiving multiple doses of the vaccine. The goal is to overcome the reduced vaccine efficacy (hypo-responsiveness to the vaccine) reported in actively or chronically infected adults.

DETAILED DESCRIPTION:
PATH and GlaxoSmithKline (GSK) are committed to developing a malaria vaccine to help reduce the burden of malaria disease in children and contribute to malaria elimination. GSK has developed a candidate vaccine against malaria caused by P. falciparum called RTS,S/AS01E. The vaccine has been shown to be safe in multiple trials and efficacy data in pediatric populations has led to a pilot implementation program in three African countries including Kenya. The RTS,S/AS01E vaccine mechanism of action is presumed to work on the initial sporozoite and liver stages of P. falciparum infection through neutralization of the circumsporozoite (CS) antigen on parasites invading after a mosquito bite in individuals immunized with the RTS,S/AS01E vaccine. In order to inform whether a vaccine such as RTS,S/AS01E may have a future role in malaria elimination, it will be important to establish vaccine efficacy in adults in Sub-Saharan Africa who are reservoirs of parasites and who contribute to ongoing malaria transmission. However, in previous trials, the vaccine has been less effective in adults who have had malaria before. There are probably multiple reasons for this, but one possible reason that is probably very important is that prior infection with malaria or an infection with malaria for long periods, even without symptoms of the disease, can prevent the vaccine from working properly.

This study postulates that treatment of infection prior to immunization can reset the immune response leading to an improved vaccine efficacy. To evaluate this hypothesis, the study will recruit 5 groups. Groups 1 and 4 will have asymptomatic infection with P. falciparum as measured by a highly sensitive polymerase chain reaction (PCR) assay and will be treated with antimalarial medications prior to immunization with RTS,S/AS01E or the comparator rabies vaccine, respectively, with the primary objective of evaluating the vaccine efficacy of RTS,S/AS01E relative to the rabies vaccine in this context. Groups 2 and 5 will be negative for asymptomatic infection with P. falciparum as measured by a highly sensitive PCR assay and will be treated with antimalarial medications prior to immunization with RTS,S/AS01E or the comparator rabies vaccine, respectively, with the secondary objective of evaluating the vaccine efficacy of RTS,S/AS01 relative to the rabies vaccine in this context. Group 3 will have asymptomatic infection with P. falciparum as measured by a highly sensitive PCR assay but will not be treated with antimalarial medications prior to immunization with the RTS,S/AS01E vaccine; the immunological profile of this group and groups 1 and 2 will be evaluated as part of secondary and exploratory objectives. Other secondary objectives include safety assessments.

The study will include an initial immunization period (vaccine given on 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations) followed by 6-12 months of follow-up (varying based on the number of events),

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed or thumb printed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female between 18 and 55 years of age, inclusive
* In good general health as evidenced by medical history and clinical examination before entering the study
* Ability to take oral medication and be willing to adhere to the medication regimen
* For females, she must be of non-childbearing potential or use appropriate measures to prevent pregnancy for 30 days prior to vaccination through 2 months after completion of the vaccine series. Non-childbearing potential means she is surgically sterilized or at least one year post-menopausal. Appropriate measures to prevent pregnancy include abstinence or adequate contraceptive precautions (i.e. intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant or Depo-Provera). Clinical trial site staff will assist with provision of acceptable birth control for study entry and will discuss with volunteer at screening visit.

Exclusion Criteria:

* Planned administration/administration of a vaccine not foreseen by the study protocol from within 30 days before the first dose of study vaccine until 30 days after the last dose of study vaccine.†

  † In the context of the COVID-19 pandemic, the administration of the COVID-19 vaccine will be allowed as an exception to this exclusion criteria as follows. The study team will work with the participant to attempt to have any COVID-19 vaccine administration occur 30 days or more before or after study vaccinations. When this is not possible, COVID-19 vaccination will be allowed 10 days or more before or after study vaccination. Intervals shorter than 10 days can be allowed on a case-by-case basis in discussion with the sponsor.
* Any prior receipt of any rabies vaccine or experimental malaria vaccine.
* Confirmed or suspected significant immunosuppressive or immunodeficient condition as determined by the investigator, including clinical stage 3 or 4 human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic reactions, significant immunoglobulin E (IgE)-mediated events or anaphylaxis to previous immunizations.
* History of any neurologic disorders.
* Acute disease (defined as the presence of a moderate or severe illness with or without fever), including acute malaria, at the time of enrolment. All vaccines can be administered to persons with a minor illness, such as diarrhea or mild upper respiratory infection without fever, i.e. Oral temperature < 37.5°C*. Individuals excluded with acute disease, including acute malaria, can become eligible again after complete recovery of the illness, including appropriate treatment as applicable, and can be rescreened at a later date. *Temperature readings may be taken by site staff either using either oral, axillary, or infrared thermal thermometers during clinic or field visits, while subjects enrolled in the reactogenicity cohort will be supplied with oral thermometers for the purposes of recording their own temperature measurements in the memory aid over 7 days after each vaccination.
* Acute or chronic, clinically significant pulmonary, cardiovascular (including cardiac arrythmias) , hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory screening tests.
* History of homozygous sickle cell disease (Hgb SS).
* Any clinically significant laboratory abnormalities as determined by the investigator on screening labs.
* History of splenectomy.
* Administration of immunoglobulins, blood transfusions or other blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant (i.e. a positive pregnancy test) or lactating female during immunization phase of the study (refer to section 2.3 for rationale). If a woman becomes pregnant after all vaccinations are complete, she will not be excluded from the remainder of the study.
* Female planning to become pregnant or planning to discontinue contraceptive precautions during the vaccination phase.
* History of chronic alcohol consumption and/or drug abuse.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose (for corticosteroids, this will mean prednisone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Major congenital defects or serious chronic illness.
* Simultaneous participation in any other clinical trial [apart from participation in the Health and Demographics Surveillance System (HDSS) network].
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 620 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O Tina, MD, MTM&H, Principal Investigator — Kombewa Clinical Research Center
Locations (1):
- Lucas O Tina, Kisumu, Kisumu County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] RTS,S Clinical Trials Partnership; Agnandji ST, Lell B, Soulanoudjingar SS, Fernandes JF, Abossolo BP, Conzelmann C, Methogo BG, Doucka Y, Flamen A, Mordmuller B, Issifou S, Kremsner PG, Sacarlal J, Aide P, Lanaspa M, Aponte JJ, Nhamuave A, Quelhas D, Bassat Q, Mandjate S, Macete E, Alonso P, Abdulla S, Salim N, Juma O, Shomari M, Shubis K, Machera F, Hamad AS, Minja R, Mtoro A, Sykes A, Ahmed S, Urassa AM, Ali AM, Mwangoka G, Tanner M, Tinto H, D'Alessandro U, Sorgho H, Valea I, Tahita MC, Kabore W, Ouedraogo S, Sandrine Y, Guiguemde RT, Ouedraogo JB, Hamel MJ, Kariuki S, Odero C, Oneko M, Otieno K, Awino N, Omoto J, Williamson J, Muturi-Kioi V, Laserson KF, Slutsker L, Otieno W, Otieno L, Nekoye O, Gondi S, Otieno A, Ogutu B, Wasuna R, Owira V, Jones D, Onyango AA, Njuguna P, Chilengi R, Akoo P, Kerubo C, Gitaka J, Maingi C, Lang T, Olotu A, Tsofa B, Bejon P, Peshu N, Marsh K, Owusu-Agyei S, Asante KP, Osei-Kwakye K, Boahen O, Ayamba S, Kayan K, Owusu-Ofori R, Dosoo D, Asante I, Adjei G, Adjei G, Chandramohan D, Greenwood B, Lusingu J, Gesase S, Malabeja A, Abdul O, Kilavo H, Mahende C, Liheluka E, Lemnge M, Theander T, Drakeley C, Ansong D, Agbenyega T, Adjei S, Boateng HO, Rettig T, Bawa J, Sylverken J, Sambian D, Agyekum A, Owusu L, Martinson F, Hoffman I, Mvalo T, Kamthunzi P, Nkomo R, Msika A, Jumbe A, Chome N, Nyakuipa D, Chintedza J, Ballou WR, Bruls M, Cohen J, Guerra Y, Jongert E, Lapierre D, Leach A, Lievens M, Ofori-Anyinam O, Vekemans J, Carter T, Leboulleux D, Loucq C, Radford A, Savarese B, Schellenberg D, Sillman M, Vansadia P. First results of phase 3 trial of RTS,S/AS01 malaria vaccine in African children. N Engl J Med. 2011 Nov 17;365(20):1863-75. doi: 10.1056/NEJMoa1102287. Epub 2011 Oct 18. PMID 22007715
- [Background] RTS,S Clinical Trials Partnership; Agnandji ST, Lell B, Fernandes JF, Abossolo BP, Methogo BG, Kabwende AL, Adegnika AA, Mordmuller B, Issifou S, Kremsner PG, Sacarlal J, Aide P, Lanaspa M, Aponte JJ, Machevo S, Acacio S, Bulo H, Sigauque B, Macete E, Alonso P, Abdulla S, Salim N, Minja R, Mpina M, Ahmed S, Ali AM, Mtoro AT, Hamad AS, Mutani P, Tanner M, Tinto H, D'Alessandro U, Sorgho H, Valea I, Bihoun B, Guiraud I, Kabore B, Sombie O, Guiguemde RT, Ouedraogo JB, Hamel MJ, Kariuki S, Oneko M, Odero C, Otieno K, Awino N, McMorrow M, Muturi-Kioi V, Laserson KF, Slutsker L, Otieno W, Otieno L, Otsyula N, Gondi S, Otieno A, Owira V, Oguk E, Odongo G, Woods JB, Ogutu B, Njuguna P, Chilengi R, Akoo P, Kerubo C, Maingi C, Lang T, Olotu A, Bejon P, Marsh K, Mwambingu G, Owusu-Agyei S, Asante KP, Osei-Kwakye K, Boahen O, Dosoo D, Asante I, Adjei G, Kwara E, Chandramohan D, Greenwood B, Lusingu J, Gesase S, Malabeja A, Abdul O, Mahende C, Liheluka E, Malle L, Lemnge M, Theander TG, Drakeley C, Ansong D, Agbenyega T, Adjei S, Boateng HO, Rettig T, Bawa J, Sylverken J, Sambian D, Sarfo A, Agyekum A, Martinson F, Hoffman I, Mvalo T, Kamthunzi P, Nkomo R, Tembo T, Tegha G, Tsidya M, Kilembe J, Chawinga C, Ballou WR, Cohen J, Guerra Y, Jongert E, Lapierre D, Leach A, Lievens M, Ofori-Anyinam O, Olivier A, Vekemans J, Carter T, Kaslow D, Leboulleux D, Loucq C, Radford A, Savarese B, Schellenberg D, Sillman M, Vansadia P. A phase 3 trial of RTS,S/AS01 malaria vaccine in African infants. N Engl J Med. 2012 Dec 13;367(24):2284-95. doi: 10.1056/NEJMoa1208394. Epub 2012 Nov 9. PMID 23136909
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of the RTS,S/AS01 malaria vaccine during 18 months after vaccination: a phase 3 randomized, controlled trial in children and young infants at 11 African sites. PLoS Med. 2014 Jul 29;11(7):e1001685. doi: 10.1371/journal.pmed.1001685. eCollection 2014 Jul. PMID 25072396
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of RTS,S/AS01 malaria vaccine with or without a booster dose in infants and children in Africa: final results of a phase 3, individually randomised, controlled trial. Lancet. 2015 Jul 4;386(9988):31-45. doi: 10.1016/S0140-6736(15)60721-8. Epub 2015 Apr 23. PMID 25913272
- [Background] Kester KE, Cummings JF, Ofori-Anyinam O, Ockenhouse CF, Krzych U, Moris P, Schwenk R, Nielsen RA, Debebe Z, Pinelis E, Juompan L, Williams J, Dowler M, Stewart VA, Wirtz RA, Dubois MC, Lievens M, Cohen J, Ballou WR, Heppner DG Jr; RTS,S Vaccine Evaluation Group. Randomized, double-blind, phase 2a trial of falciparum malaria vaccines RTS,S/AS01B and RTS,S/AS02A in malaria-naive adults: safety, efficacy, and immunologic associates of protection. J Infect Dis. 2009 Aug 1;200(3):337-46. doi: 10.1086/600120. PMID 19569965
- [Background] Regules JA, Cicatelli SB, Bennett JW, Paolino KM, Twomey PS, Moon JE, Kathcart AK, Hauns KD, Komisar JL, Qabar AN, Davidson SA, Dutta S, Griffith ME, Magee CD, Wojnarski M, Livezey JR, Kress AT, Waterman PE, Jongert E, Wille-Reece U, Volkmuth W, Emerling D, Robinson WH, Lievens M, Morelle D, Lee CK, Yassin-Rajkumar B, Weltzin R, Cohen J, Paris RM, Waters NC, Birkett AJ, Kaslow DC, Ballou WR, Ockenhouse CF, Vekemans J. Fractional Third and Fourth Dose of RTS,S/AS01 Malaria Candidate Vaccine: A Phase 2a Controlled Human Malaria Parasite Infection and Immunogenicity Study. J Infect Dis. 2016 Sep 1;214(5):762-71. doi: 10.1093/infdis/jiw237. Epub 2016 Jun 13. PMID 27296848
- [Background] Moorthy VS, Ballou WR. Immunological mechanisms underlying protection mediated by RTS,S: a review of the available data. Malar J. 2009 Dec 30;8:312. doi: 10.1186/1475-2875-8-312. PMID 20042088
- [Background] Polhemus ME, Remich SA, Ogutu BR, Waitumbi JN, Otieno L, Apollo S, Cummings JF, Kester KE, Ockenhouse CF, Stewart A, Ofori-Anyinam O, Ramboer I, Cahill CP, Lievens M, Dubois MC, Demoitie MA, Leach A, Cohen J, Ballou WR, Heppner DG Jr. Evaluation of RTS,S/AS02A and RTS,S/AS01B in adults in a high malaria transmission area. PLoS One. 2009 Jul 31;4(7):e6465. doi: 10.1371/journal.pone.0006465. PMID 19649245
- [Background] Wykes MN, Horne-Debets JM, Leow CY, Karunarathne DS. Malaria drives T cells to exhaustion. Front Microbiol. 2014 May 27;5:249. doi: 10.3389/fmicb.2014.00249. eCollection 2014. PMID 24904561
- [Background] Keitany GJ, Kim KS, Krishnamurty AT, Hondowicz BD, Hahn WO, Dambrauskas N, Sather DN, Vaughan AM, Kappe SHI, Pepper M. Blood Stage Malaria Disrupts Humoral Immunity to the Pre-erythrocytic Stage Circumsporozoite Protein. Cell Rep. 2016 Dec 20;17(12):3193-3205. doi: 10.1016/j.celrep.2016.11.060. PMID 28009289
- [Background] Illingworth J, Butler NS, Roetynck S, Mwacharo J, Pierce SK, Bejon P, Crompton PD, Marsh K, Ndungu FM. Chronic exposure to Plasmodium falciparum is associated with phenotypic evidence of B and T cell exhaustion. J Immunol. 2013 Feb 1;190(3):1038-47. doi: 10.4049/jimmunol.1202438. Epub 2012 Dec 21. PMID 23264654
- [Background] Freeman GJ, Sharpe AH. A new therapeutic strategy for malaria: targeting T cell exhaustion. Nat Immunol. 2012 Jan 19;13(2):113-5. doi: 10.1038/ni.2211. PMID 22261959
- [Background] Weiss GE, Crompton PD, Li S, Walsh LA, Moir S, Traore B, Kayentao K, Ongoiba A, Doumbo OK, Pierce SK. Atypical memory B cells are greatly expanded in individuals living in a malaria-endemic area. J Immunol. 2009 Aug 1;183(3):2176-82. doi: 10.4049/jimmunol.0901297. Epub 2009 Jul 10. PMID 19592645
- [Background] Weiss GE, Traore B, Kayentao K, Ongoiba A, Doumbo S, Doumtabe D, Kone Y, Dia S, Guindo A, Traore A, Huang CY, Miura K, Mircetic M, Li S, Baughman A, Narum DL, Miller LH, Doumbo OK, Pierce SK, Crompton PD. The Plasmodium falciparum-specific human memory B cell compartment expands gradually with repeated malaria infections. PLoS Pathog. 2010 May 20;6(5):e1000912. doi: 10.1371/journal.ppat.1000912. PMID 20502681
- [Background] Butler NS, Moebius J, Pewe LL, Traore B, Doumbo OK, Tygrett LT, Waldschmidt TJ, Crompton PD, Harty JT. Therapeutic blockade of PD-L1 and LAG-3 rapidly clears established blood-stage Plasmodium infection. Nat Immunol. 2011 Dec 11;13(2):188-95. doi: 10.1038/ni.2180. PMID 22157630
- [Background] Nielsen CM, Vekemans J, Lievens M, Kester KE, Regules JA, Ockenhouse CF. RTS,S malaria vaccine efficacy and immunogenicity during Plasmodium falciparum challenge is associated with HLA genotype. Vaccine. 2018 Mar 14;36(12):1637-1642. doi: 10.1016/j.vaccine.2018.01.069. Epub 2018 Feb 10. PMID 29439870
- [Derived] Copeland NK, Otieno L, Otieno JD, Otieno S, Chira S, Ivinson K, Onyango I, Wasuna R, Akala H, Onditi A, Sifuna P, Andagalu B, Oyugi R, Omondi M, Amoit S, Locke E, Gregory S, Bergmann-Leitner ES, Pindolia H, Raine M, Gast C, Mercer LD, Aponte JJ, Lievens M, Ockenhouse CF, Lee CK. Efficacy of RTS,S/AS01E Only Seen in Baseline Parasitemic and Not Baseline Aparasitemic Plasmodium falciparum-Exposed, Drug-Treated Kenyan Adults. J Infect Dis. 2025 Sep 15;232(3):e372-e382. doi: 10.1093/infdis/jiaf274. PMID 40439411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the villages in the Kombewa Health and Demographics Surveillance System (HDSS) consisting of half of Kisumu West and all of Seme sub-counties of Kisumu County, Kenya.
  Prior to enrollment participants were tested for the presence or absence of asymptomatic infection with Plasmodium falciparum (P. falciparum, the parasite that causes malaria) measured using a highly sensitive polymerase chain reaction (PCR) assay.
Pre-assignment Details: Participants were stratified by baseline P. falciparum parasitemia status and then block randomized. The first 105 participants who were positive for parasitemia at baseline were randomized in a 1:1:1 ratio with 35 participants assigned to each of Groups 1, 3 and 4. The next 258 participants with baseline parasitemia were randomized in a 1:1 ratio to Groups 1 and 4. Participants who were negative for parasitemia at baseline were randomized in a 1:1 ratio to Groups 2 and 5.
Groups:
- Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine: Participants with detectable Plasmodium falciparum parasitemia at baseline received anti-malarial treatment with dihydroartemisinin-piperaquine (DHA/Pip) plus low dose primaquine (LD PQ) 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a course of artemether/lumefantrine (A/L) plus LD PQ was administered.
  Participants were randomized to receive 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
- Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine: Participants with no detectable P. falciparum parasitemia at baseline received anti-malarial prophylaxis with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and a 2nd course of DHA/Pip plus LD PQ 2 weeks before the second vaccination. One week before the third vaccination, a course of A/L plus LD PQ was administered.
  Participants were randomized to receive 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
- Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine: Participants with detectable P. falciparum parasitemia at baseline did not receive any anti-malarial medications to clear parasites.
  Participants were randomized to receive 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
  This group is included only for immunological assessment and not for vaccine efficacy.
- Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine: Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with dihydroartemisinin-piperaquine (DHA/Pip) plus low dose primaquine (LD PQ) 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a three-day course of artemether/lumefantrine (A/L) plus LD PQ was administered.
  Participants were randomized to receive 3 vaccinations of Abhayrab rabies vaccine on a 0, 1, 7 month schedule.
- Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine: Participants with no detectable P. falciparum parasitemia at baseline received anti-malarial prophylaxis with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and a 2nd course of DHA/Pip plus LD PQ 2 weeks before the second vaccination. One week before the third vaccination, a course of A/L plus LD PQ was administered.
  Participants were randomized to receive 3 vaccinations of Abhayrab rabies vaccine on a 0, 1, 7 month schedule.
Period: Overall Study
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Started | 164 | 128 | 36 | 164 | 128
Received Study Vaccination | 160 | 124 | 35 | 159 | 127
Completed | 136 | 108 | 32 | 148 | 115
Not Completed | 28 | 20 | 4 | 16 | 13
Not completed — Lost to Follow-up | 19 | 10 | 2 | 7 | 11
Not completed — Physician Decision | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 1 | 1 | 1
Not completed — Randomized but Did Not Receive Study Product | 4 | 4 | 1 | 5 | 1

BASELINE CHARACTERISTICS:
Population: The total vaccinated cohort (TVC) includes all randomized participants who received at least one vaccination.
Groups:
- Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine: Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a course of A/L plus LD PQ was administered.
  Participants were randomized to receive 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
- Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine: Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a three-day course of A/L plus LD PQ was administered.
  Participants were randomized to receive 3 vaccinations of Abhayrab rabies vaccine on a 0, 1, 7 month schedule.
- Total: Total of all reporting groups
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine | Total
Number analyzed (Participants) | 160 | 124 | 35 | 159 | 127 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.94 (8.04) | 34.02 (7.63) | 34.57 (8.93) | 31.76 (8.49) | 34.04 (8.04) | 32.91 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 80 | 21 | 75 | 75 | 323
  Male | 88 | 44 | 14 | 84 | 52 | 282
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 160 | 124 | 35 | 159 | 127 | 605
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Luo | 158 | 122 | 35 | 159 | 125 | 599
  Luhya | 2 | 2 | 0 | 0 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Kenya | 160 | 124 | 35 | 159 | 127 | 605

OUTCOME MEASURES:

1. Primary Outcome: Time to First PCR-detectable Malaria Infection During the Active Detection of Infection (ADI) Phase in Groups 1 and 4
Description: Participants were actively monitored for malarial infection starting 2 weeks after the third vaccination. Blood samples were assayed using a highly sensitive polymerase chain reaction (PCR) (Plasmodium falciparum/ Pan-Plasmodium 18S ribosomal ribonucleic acid (rRNA) laboratory developed test [LDT]) that can detect sub-clinical parasitemia at the US Army Medical Research Directorate-Africa (USAMRD-A) / Kenya Medical Research Institute (KEMRI) laboratories in Kisumu, Kenya. A positive PCR result from blood samples collected during the ADI was recorded as a positive event for the presence of P. falciparum blood stage infection.
  The time to first malaria infection is expressed in terms of rate of first malaria infection, that is, the number of malaria infection events reported over the time period elapsed until the event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group.
Time Frame: The active detection of infection phase began 2 weeks after the third vaccination (approximately week 30) for up to 35 weeks. Participants provided blood samples every 21 days during the ADI phase for PCR assays.
Population: The primary endpoint was pre-specified to be analyzed in Groups 1 and 4 only. The According to Protocol (ATP) cohort for efficacy includes all participants in the TVC with no major protocol deviations that could potentially interfere with the efficacy assessment of the study vaccine and who contributed to the time at risk starting 14 days after the third dose.
Measure: Number; unit: Events per person year at risk
Groups:
- Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine: Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a course of A/L plus LD PQ was administered.
  Participants received 3 vaccinations with malarial vaccine RTS,S/AS01E by intramuscular injection given on a 0, 1, and 7 month schedule with the final dose being 1/5 of the dose of the first two immunizations.
- Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine: Participants with detectable P. falciparum parasitemia at baseline received anti-malarial treatment with DHA/Pip plus LD PQ 4 weeks prior to the first vaccination and another course of DHA/Pip plus LD PQ two weeks before the second vaccination. One week before the third vaccination, a three-day course of A/L plus LD PQ was administered.
  Participants received 3 vaccinations of Abhayrab rabies vaccine on a 0, 1, 7 month schedule.
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine
Number analyzed (Participants) | 151 | 151
Events per person year at risk | 1.01 | 1.49
Statistical Analysis 1: Comparison: Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine vs Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine; Vaccine efficacy against the first PCR-positive P. falciparum infection among adults who were P. falciparum positive at baseline was assessed using Cox proportional hazards regression model with a covariate for group assignment to compare Groups 1 and 4. HIV status, Age (tertiles), and sleep under a bednet were included as covariates; Test type: Other; p = 0.009, Wald test; Vaccine Efficacy = 35.9, 95% CI 2-sided [10.3 to 54.2] — Vaccine efficacy (VE) is defined as the percent reduction in the hazard, i.e. one minus the hazard ratio (HR, RTS,S/AS01E Vaccine vs. Rabies vaccine)

2. Secondary Outcome: Time to First PCR-detectable Malaria Infection During the Active Detection of Infection Phase in Groups 2 and 5
Description: Participants were actively monitored for malarial infection starting 2 weeks after the third vaccination. Blood samples were assayed using a highly sensitive PCR (Plasmodium falciparum/ Pan-Plasmodium 18S rRNA LDT) that can detect sub-clinical parasitemia. A positive PCR result from blood samples collected during the ADI phase was recorded as a positive event for the presence of P. falciparum blood stage infection.
  The time to first malaria infection is expressed in terms of rate of first malaria infection, that is, the number of malaria infection events reported over the time period elapsed until the event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group.
Time Frame: as for outcome 1
Population: This endpoint was pre-specified to be analyzed in Groups 2 and 5 only. The ATP cohort for efficacy includes all participants in the TVC with no major protocol deviations that could potentially interfere with the efficacy assessment of the study vaccine and who contributed to the time at risk starting 14 days after the third dose.
Measure: Number; unit: Events per person year at risk
Arm/Group | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Number analyzed (Participants) | 118 | 123
Events per person year at risk | 0.77 | 0.62
Statistical Analysis 1: Comparison: Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine vs Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine; Vaccine efficacy against the first PCR-positive P. falciparum infection among adults who were P. falciparum positive at baseline was assessed using Cox proportional hazards regression model with a covariate for group assignment to compare Groups 2 and 5. HIV status, Age (tertiles), and sleep under a bednet were included as covariates; Test type: Other; p = 0.369, Wald test; Vaccine Efficacy = -24, 95% CI 2-sided [-97 to 22.2] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, or temporally associated with a study procedure.
  A serious adverse event is any adverse event that:
  * Resulted in death,
  * Was life-threatening,
  * Resulted in disability/incapacity,
  * Required hospitalization or prolongation of existing hospitalization,
  * Resulted in disability/incapacity.
  * Resulted in a congenital anomaly and / or birth defect.
Time Frame: From first dose to end of study, up to 65 weeks.
Population: The Safety analysis population includes all enrolled participants who received at least one vaccination and for whom any safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Number analyzed (Participants) | 160 | 124 | 35 | 159 | 127
Participants | 3 | 2 | 1 | 1 | 3

4. Secondary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AEs)
Description: Solicited AEs are pre-specified local and systemic AEs that occur relatively more frequently or are known to be associated with immunization, which are monitored actively as potential indicators of vaccine reactogenicity.
  Solicited local and general AEs were collected among RTS,S vaccinated groups in the first 50 participants enrolled in Groups 1 and 2 and all participants enrolled in Group 3 (Reactogenicity Cohort) for seven days (day of vaccination and six subsequent days) after each dose of vaccine.
  Local (injection site) adverse events are defined as:
  * Pain at injection site
  * Swelling at injection site
  Systemic adverse events are defined as:
  * Fever (temperature ≥ 37.5°C)
  * Headache
  * Gastrointestinal problems
  * Fatigue
  * Muscle ache
Time Frame: Within 7 days after each vaccination.
Population: The Reactogenicity Cohort (the first 50 participants in Groups 1 and 2 and all participants in Group 3) with available reactogenicity data.
  Participants in Groups 4 and 5 did not have solicited AEs collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Number analyzed (Participants) | 49 | 47 | 35 | 0 | 0
Participants
  Local Solicited AEs | 24 | 26 | 14 |  |
  Systemic Solicited AEs | 20 | 16 | 14 |  |

5. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, or temporally associated with a study procedure.
  Unsolicited AEs are any AEs reported spontaneously by the participant, observed by the study staff during study visits or those identified during review of medical records or source documents. Solicited AEs with an onset after the seven-day solicitation period were also considered unsolicited AEs.
Time Frame: Within 28 days after each vaccination.
Population: All enrolled participants who received at least one vaccination and for whom any safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
Number analyzed (Participants) | 160 | 124 | 35 | 159 | 127
Participants | 103 | 87 | 20 | 110 | 92

6. Secondary Outcome: Geometric Mean Titer of Anti-Plasmodium Falciparum Circumsporozoite (CS) Antibodies in Groups 1, 2, and 3
Description: The RTS,S antigen consists of sequences of both the P. falciparum circumsporozoite protein and hepatitis B surface antigen.
  Antibody levels against P. falciparum circumsporozoite (CS) protein central repeat region (NANP) were measured from blood samples of participants in Groups 1, 2 and 3 using standard enzyme-linked immunosorbent assays (ELISA) at Walter Reed Army Institute of Research (WRAIR), in Silver Spring, MD, United States.
Time Frame: Baseline, Day 29 (28 days after first vaccination), Day 57 (28 days after second vaccination), Day 197 (24 weeks after second vaccination), and Day 225 (28 days after third vaccination)
Population: The ATP cohort for immunogenicity included all participants in the TVC who received all vaccinations according to protocol procedures and within the protocol specified intervals, performed blood samplings for immunogenicity according to protocol intervals, and did not use any medication or blood products forbidden by the protocol and did not have any reported underlying medical condition influencing immune responses. Participants with available data at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine
Number analyzed (Participants) | 151 | 118 | 34
titer
  Baseline | 171.89 [139.82 to 211.33] | 139.80 [110.54 to 176.80] | 231.64 [144.16 to 372.21]
  Day 29 | 2328.78 [1922.14 to 2821.44] | 2538.76 [2057.52 to 3132.57] | 2744.34 [1809.21 to 4162.80]
  Day 57: number analyzed (Participants) | 151 | 117 | 34
  Day 57 | 3391.18 [2887.17 to 3983.18] | 3530.57 [2986.65 to 4173.54] | 4708.33 [3342.96 to 6631.36]
  Day 197 | 1627.01 [1381.90 to 1915.59] | 1584.13 [1343.47 to 1867.90] | 1751.77 [1229.91 to 2495.05]
  Day 225: number analyzed (Participants) | 150 | 118 | 34
  Day 225 | 2121.04 [1803.76 to 2494.12] | 2519.28 [2132.57 to 2976.12] | 2586.04 [1864.68 to 3586.46]

7. Secondary Outcome: Anti-Plasmodium Falciparum Circumsporozoite (CS) Antibody Avidity Index in Groups 1, 2, and 3
Description: Antibody levels against P. falciparum circumsporozoite (CS) protein central repeat region (NANP) measured by standard enzyme-linked immunosorbent assays (ELISA) for participants in Groups 1, 2 and 3. To measure antibody-antigen avidity (strength of binding) ELISA was performed with and without urea (to dissociate the antigen-antibody complex).
  The avidity index is calculated by dividing the serum titer obtained in the presence of the urea by the serum titer without urea.
Time Frame: as for outcome 6
Population: The according to protocol (ATP) cohort for immunogenicity; participants with available data at each time point.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine
Number analyzed (Participants) | 151 | 118 | 34
ratio
  Baseline | 0.62 [0.58 to 0.65] | 0.64 [0.60 to 0.68] | 0.65 [0.57 to 0.73]
  Day 29 | 0.64 [0.62 to 0.67] | 0.67 [0.65 to 0.70] | 0.69 [0.62 to 0.76]
  Day 57: number analyzed (Participants) | 151 | 117 | 34
  Day 57 | 0.63 [0.60 to 0.65] | 0.64 [0.61 to 0.67] | 0.67 [0.62 to 0.72]
  Day 197 | 0.59 [0.57 to 0.62] | 0.63 [0.60 to 0.66] | 0.66 [0.60 to 0.71]
  Day 225: number analyzed (Participants) | 150 | 118 | 34
  Day 225 | 0.55 [0.53 to 0.58] | 0.65 [0.62 to 0.68] | 0.66 [0.60 to 0.72]

8. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-Hepatitis B Surface Antigen (HBsAg) Antibodies in Groups 1, 2, and 3
Description: The RTS,S vaccine antigen consists of sequences of both the P. falciparum circumsporozoite protein and hepatitis B surface antigen, hence anti-HBsAg antibodies were also measured.
  Anti-hepatitis B surface antigen antibodies were assessed at the International AIDS Vaccine Initiative Human Immunology Laboratory (IAVI-HIL) at Imperial College, London, UK, using a commercially available ELISA kit.
Time Frame: Baseline, Day 29 (28 days after first vaccination) and Day 225 (28 days after third vaccination)
Population: ATP Cohort for Immunogenicity with available data at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine
Number analyzed (Participants) | 151 | 118 | 34
titer
  Baseline | 16.88 [12.56 to 22.69] | 14.32 [10.25 to 19.99] | 15.57 [8.47 to 28.63]
  Day 29 | 61.27 [36.80 to 102.00] | 60.16 [34.48 to 104.96] | 87.89 [23.73 to 325.44]
  Day 225: number analyzed (Participants) | 150 | 118 | 34
  Day 225 | 1500.56 [1014.34 to 2219.85] | 1789.89 [1237.46 to 2588.91] | 2321.30 [1255.51 to 4291.81]

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events are reported through the end of the study, up to 65 weeks Non-serious adverse events were collected up to 28 days following administration of each dose of vaccine and, where applicable, course of per protocol scheduled anti-malarial treatment.
Description: All-cause mortality is reported for all randomized participants. Adverse events are reported for all participants who received at least one vaccination.
Arm/Group | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine
All-Cause Mortality (participants affected / at risk) | 1/164 | 0/128 | 0/36 | 0/164 | 0/128
Serious Adverse Events (participants affected / at risk) | 3/160 | 2/124 | 1/35 | 1/159 | 3/127
Other Adverse Events (participants affected / at risk) | 111/160 | 96/124 | 25/35 | 110/159 | 92/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine (N=160) | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine (N=124) | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine (N=35) | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine (N=159) | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine (N=127)
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyomyositis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Alcoholic coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Positive Parasitemia; Anti-malarial Treatment + RTS,S/AS01E Vaccine (N=160) | Group 2: No Parasitemia; Anti-malarial Prophylaxis + RTS,S/AS01E Vaccine (N=124) | Group 3: Positive Parasitemia; RTS,S/AS01E Vaccine (N=35) | Group 4: Positive Parasitemia; Anti-malarial Treatment + Rabies Vaccine (N=159) | Group 5: No Parasitemia, Anti-malarial Prophylaxis + Rabies Vaccine (N=127)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 2 | 2 | 0 | 1 | 2
Myopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 1 | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 2 | 5 | 0 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Epulis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 5 | 5 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 5 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 10 | 10 | 8 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 24 | 25 | 14 | 0 | 0
Injection site swelling (General disorders) | 7 | 10 | 5 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 4 | 2 | 3 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Bartholin's abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Body tinea (Infections and infestations) | 4 | 4 | 2 | 5 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 7 | 1 | 0 | 3 | 2
Conjunctivitis (Immune system disorders) | 5 | 9 | 1 | 2 | 7
Dermatitis infected (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 1 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 2 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Malaria (Infections and infestations) | 15 | 15 | 5 | 19 | 16
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 2 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 2 | 1 | 0 | 3 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 2 | 4
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 24 | 10 | 4 | 39 | 22
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Schistosomiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Septic rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sexually transmitted disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tinea capitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 2 | 1 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 3 | 3 | 0 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 18 | 0 | 19 | 16
Urethritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 5 | 0 | 2 | 3
Vulvovaginal candidiasis (Infections and infestations) | 1 | 2 | 1 | 2 | 4
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 5 | 4 | 1 | 4 | 3
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 9 | 0 | 14 | 9
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 15 | 7 | 9 | 8
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 24 | 18 | 9 | 14 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT04661579/Prot_001.pdf
  • Statistical Analysis Plan (2023-04-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04661579/SAP_002.pdf
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04661579/ICF_000.pdf